CLINICAL TRIAL: NCT04287660
Title: A Phase 3, Single Arm, Multi-Center Study to Assess the Efficacy and Safety of Clarithromycin(Biaxin)-Lenalidomide-Low-Dose-Dexamethasone (BiRd) Combined With B-cell Maturation Antigen (BCMA)-Directed Chimeric Antigen Receptor (CAR) T-cell Therapy in Patients With Newly Diagnosed Multiple Myeloma
Brief Title: Study of BiRd Regimen Combined With BCMA CAR T-cell Therapy in Newly Diagnosed Multiple Myeloma (MM) Patients
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Collaborators: Changshu Frist People's Hospital (Unknown); The Second People's Hospital of Huai'an (Other); Affiliated Hospital of Jiangnan University (Other); Jiangsu Province Hospital of Traditional Chinese Medicine (Other); Jiangyin People's Hospital (Other); Jingjiang People's Hospital (Other); The Third People's Hospital of Kunshan (Unknown); Lianyungang Hospital Affiliated Bengbu Medical College (Other); Suzhou Municipal Hospital (Other); Zhangjiagang First People's Hospital (Other); Shanghai Unicar-Therapy Bio-medicine Technology Co.,Ltd (Industry); The First Affiliated Hospital with Nanjing Medical University (Other); Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BiRd-01
Record Dates: First submitted 2020-02-19; First posted 2020-02-27 (Actual); Last update posted 2021-10-25 (Actual); Status verified 2021-02

CONDITIONS: Multiple Myeloma
Keywords: BiRd; CART; BCMA; MM
MeSH Terms: conditions — Multiple Myeloma | interventions — Clarithromycin; Lenalidomide; Dexamethasone

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BiRd combined with BCMA CAR T-cells infusion (Experimental)
  Interventions: Drug: clarithromycin, lenalidomide, dexamethasone and autologous BCMA-directed CAR T-cells

INTERVENTIONS:
Drug: clarithromycin, lenalidomide, dexamethasone and autologous BCMA-directed CAR T-cells — * clarithromycin: 500mg, PO, twice daily, on days 1~21 for a 28-day cycle.
  * lenalidomide: 25mg, PO, on days 1~21 for a 28-day cycle. dexamethasone: 40mg, PO on days 1,8,15 and 22 for a 28-day cycle. BCMA CAR T cell: (2-3)×10E7/kg, intravenously infusion.
  * Doses should be adjusted according to renal function.

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of BiRd regimen combined with BCMA CAR T cell therapy in newly diagnosed multiple myeloma patients

DETAILED DESCRIPTION:
This is a phase 3, single arm, multi-center study. The patients will receive BiRd regimen (clarithromycin,lenalidomide, dexamethasone) combined with infusion of autologous BCMA-directed CAR T-cells in newly diagnosed MM patients. The study participation will be 4 years including treatment and follow-up periods.

ELIGIBILITY:
Inclusion Criteria:

1. Newly diagnosed MM according to the criteria by International Myeloma Working Group (IMWG)
2. Age 18-75
3. Eastern Cooperative Oncology Group (ECOG) score 0-2
4. BCMA positive as detected with flowcytometry or ELISA.
5. Patients with left ventricular ejection fraction ≥ 0.5 by echocardiography or grade I/II cardiovascular dysfunction according to the New York Heart Association Classification.
6. Patients with aspartate aminotransferase or glutamic-pyruvic transaminase > 3x upper limit of normal or bilirubin > 2.0 mg/dL

Exclusion Criteria:

1. Patients are pregnant or lactating.
2. Nonsecretory MM.
3. History of previous treatment of MM.
4. Patients with uncontrolled active infection.
5. Patients with active hepatitis B or hepatitis C infection.
6. Patients with HIV infection.
7. Patients with atrial or venous thrombosis or embolism.
8. Patients with myo-infarction or severe arrythmia in the recent 6 months.
9. Other comorbidities that investigators considered not suitable for this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-10-19 (Actual); Primary Completion 2023-01-31 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) | 4 weeks after CAR T-cells infusion (up to 14 weeks)
  ORR includes stringent complete response (sCR), complete remission (CR), very good partial remission (VGPR) and partial remission (PR). Stringent complete response (sCR): complete response as defined below plus normal free light chain (FLC) and absence of clonal cells in bone marrow biopsy by immunohistochemistry (κ/λ ratio ≤4:1 or ≥1:2 for κ and λ patients, respectively, after counting ≥100 plasma cells). Complete Response (CR)：negative immunofixation on the serum and urine and disappearance of any soft tissue plasmacytomas and <5% plasma cells in bone marrow aspirates. Very good partial response (VGPR)：serum and urine M-protein detectable by immunofixation but not on electrophoresis or ≥90% reduction in serum M-protein plus urine M-protein level <100 mg per 24 h. Partial response (PR): ≥50% reduction of serum M-protein plus reduction in 24 h urine M-protein by ≥90% or to <200 mg per 24 h.

SECONDARY OUTCOMES:
Overall survival (OS) | 4 years
  time from enrollment to the date of death from any cause
Event-free survival (EFS) | 4 years
  time from enrollment to the date of primary refractory disease, or relapse from sCR, or CR, or death from any cause
Cumulative incidence of relapse(CIR) | 4 years
  time from the date of achievement of a remission until the date of relapse
Number of adverse events | 2 years
  adverse events are evaluated with CTCAE V5.0

CONTACTS AND LOCATIONS:
Overall Officials: Xiaowen Tang, Ph.D, Principal Investigator — The First Affiliated Hospital of Soochow University
Locations (1):
- The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China